CLINICAL TRIAL: NCT01679587
Title: Multicenter, Randomized, Single-blind, Placebo-controlled, Combined 2-fold Cross-over and Group-comparison, Dose-escalation Study to Investigate Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Single Oral Doses of BAY 85-3934 in Subjects With Chronic Kidney Disease (CKD)
Brief Title: Dose Escalation Study to Investigate Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of BAY85-3934 in Subjects With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 16370; 2012-002375-33 (EudraCT Number)
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — molidustat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Molidustat, 80 mg (Experimental): Subjects received a single oral dose of 80 mg BAY 85-3934 in the first period and placebo in the second period, separated by a wash-out period of at least 1 week.
  Interventions: Drug: Molidustat (BAY85-3934); Drug: Placebo
- Molidustat, 120 mg (Experimental): Subjects received a single oral dose of 120 mg BAY 85-3934 in the first period and placebo in the second period, separated by a wash-out period of at least 1 week.
  Interventions: Drug: Molidustat (BAY85-3934); Drug: Placebo
- Molidustat, 40 mg (Experimental): Subjects received a single oral dose of 40 mg BAY 85-3934 in the first period and placebo in the second period, separated by a wash-out period of at least 1 week. This is an optional dose escalation step.
  Interventions: Drug: Molidustat (BAY85-3934); Drug: Placebo
- Molidustat, 160 mg (Experimental): Subjects received a single oral dose of 160 mg BAY 85-3934 in the first period and placebo in the second period, separated by a wash-out period of at least 1 week. This is an optional dose escalation step.
  Interventions: Drug: Molidustat (BAY85-3934); Drug: Placebo

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — 20 mg molidustat as a single tablet
Drug: Placebo — Single oral dose of matching placebo will be given in each treatment arm

SUMMARY:
Primary objective was to assess in subjects with CKD: Safety and tolerability of molidustat (BAY 85-3934), effects of molidustat on non-invasive hemodynamics Secondary objectives were to assess: Effects on pharmacodynamic parameters of erythropoiesis (erythropoietin, reticulocytes, erythrocytes, hemoglobin, hematocrit), pharmacokinetics of molidustat, exploratory biomarkers, ie, midregional pro-atrial natriuretic peptide, midregional pro-adrenomedullin, plasma renin activity, and optionally B-type natriuretic peptide, vascular endothelial growth factor, cyclic guanosine monophosphate, cyclic adenosine monophosphate, and noradrenaline

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic kidney disease (CKD) not on dialysis assessed by medical history and eGFR (MDRD) = < 60 mL/min estimated at the pre-study visit
* Stable renal disease, ie not expected to begin dialysis during the study
* Systolic blood pressure =>110 mmHg and =<160 mmHg
* Heart rate =<100 BPM
* Hemoglobin = >9 g/dL
* Female subjects without child-bearing potential, ie postmenopausal women with 12 months of spontaneous amenorrhea or with 6 months of spontaneous amenorrhea and serum FSH levels >30 mIU/mL, women with 6 weeks post bilateral ovariectomy, women with bilateral tubal ligation, and women with hysterectomy
* Body mass index (BMI): = >18 and = < 35 kg/m2 at the pre-study visit

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which a relevant impairment of absorption, distribution, metabolism, elimination or effects of the study drug is assumed
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Chronic heart failure, New York Heart Association (NYHA) III-IV
* Coronary artery disease with uncured significant stenosis
* Angina pectoris
* Significant stenosis of cerebral vessels
* Significant uncorrected rhythm or conduction disturbances such as a second- or third-degree atrioventricular block without a cardiac pacemaker or episodes of sustained ventricular tachycardia
* Subjects with impaired liver function (Child Pugh B to C based on medical history)
* History of thrombotic or thromboembolic events (eg myocardial infarction, stroke, transient ischemic attack, deep vein thrombosis, pulmonary embolism) within the recent 6 months
* Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy that required or is likely to require treatment (intraocular injections or laser photocoagulation) during the study
* Subjects with a history of malignant disease during the last 5 years
* Treatment with EPO-stimulating agents (ESA) or rhEPO within the last 2 weeks before first intake of study drug
* Suspicion of drug or alcohol abuse
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV 1+2) at the pre-study visit

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Approximately 9 weeks
Blood pressure | Approximately 9 weeks
  Systolic, diastolic, mean blood pressure
Heart rate | Approximately 9 weeks
Cmax | Pre-dose and up to 48 h post-dose
  Maximum observed drug concentration in measured matrix after single dose administration
Cmax/D | Pre-dose and up to 48 h post-dose
  Cmax divided by dose
AUC | Pre-dose and up to 48 h post-dose
  Area under the concentration vs time curve from zero to infinity after single dose
AUC/D | Pre-dose and up to 48 h post-dose
  AUC divided by dose
Heart rate over 1 min | Pre-dose and up to 24 h post-dose
Standing blood pressure procedure | Starting from 2 h post-dose and up to 4 h post-dose
Impedance cardiography | Pre-dose and up tp 8 h post-dose
  Stroke volume, heart rate, cardiac index, cardiac output, and total peripheral resistance

SECONDARY OUTCOMES:
Change of hematology profile | From baseline to Day 1 after single dose
  Hematology profile includes blood concentration of erythropoietin, reticulocytes, erythrocytes, hemoglobin, hematocrit, and exploratory biomarkers.
Cmax,norm | Pre-dose and up to 48 h post-dose
  Cmax divided by dose per body weight
AUCnorm | Pre-dose and up to 48 h post-dose
  AUC divided by dose per body weight
AUC(0-24) | Pre-dose and up to 24 h post-dose
  AUC from 0 until 24 h after study drug administration
AUC(0-tlast) | Pre-dose and up to 48 h post-dose
  AUC from time 0 to the last data point > lower limit of quantification
t½ | Pre-dose and up to 48 h post-dose
  Half-life associated with the terminal slope
tmax | Pre-dose and up to 48 h post-dose
  Time to reach Cmax (in case of two identical Cmax values, the first tmax was used)
MRT | Pre-dose and up to 48 h post-dose
  Mean residence time
CL/F | Pre-dose and up to 48 h post-dose
  Total body clearance of drug calculated after extravascular administration (eg, apparent oral clearance)
Vz/F | Pre-dose and up to 48 h post-dose
  Apparent volume of distribution during terminal phase after extravascular administration
Geometric mean erythropoietin Cmax | Pre-dose and up to 24 h post-dose
Geometric mean reticulocyte count | Pre-dose and up to 24 h post-dose
Geometric mean erythrocyte count | Pre-dose and up to 24 h post-dose
Geometric mean reticulocytes/erythrocytes values | Pre-dose and up to 24 h post-dose
Geometric mean hemoglobin values | Pre-dose and up to 24 h post-dose
Geometric mean hematocrit | Pre-dose and up to 24 h post-dose
Geometric mean erythropoietin tmax | Pre-dose and up to 24 h post-dose
Geometric mean erythropoietin AUC(0-24) | Pre-dose and up to 24 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Germany (3):
  - München, Bavaria
  - Mönchengladbach, North Rhine-Westphalia
  - Kiel, Schleswig-Holstein

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/